CLINICAL TRIAL: NCT01787214
Title: The Effect of Walnuts on Glucose Variability in Adults With Type-2 Diabetes Mellitus: a Dose-response Metabolic Feeding Study
Brief Title: Walnuts and Glucose Variability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Loma Linda University (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Michelle Wien, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: walnuts and glucose
Record Dates: First submitted 2013-02-01; First posted 2013-02-08 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Type-2 Diabetes
Keywords: glucose variability; glycemia; type-2 diabetes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full dose (Active Comparator): full dose of walnuts (20% energy needs)
  Interventions: Dietary Supplement: Full dose
- Half-dose (Active Comparator): Half dose of walnuts (10% of energy needs)
  Interventions: Dietary Supplement: Half dose
- Control (Other): Walnut free meals
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Full dose — 20% of daily energy needs supplied by walnuts
  Arms: Full dose
Dietary Supplement: Half dose — 10% of daily energy needs supplied by walnuts
  Arms: Half-dose
Dietary Supplement: Control — Walnut free meals
  Arms: Control

SUMMARY:
Persons with type 2 diabetes mellitus (T2DM) have swings in their blood sugar levels that may lead to a higher risk of developing heart disease. An important part of diabetes management involves eating a diet to prevent large swings in blood sugar levels. Walnuts contain fat, protein and fiber that may reduce the swings in blood sugar. The purpose of this study is to compare the effects of a walnut-free American Diabetes Association (ADA) diet versus 2 levels of walnut-enriched ADA diets on blood sugar swings. Eighteen male and female adults with T2DM will participate in the study. Subjects will be randomized to consume an ADA diet with or without walnuts for 3 consecutive days every other week. Subjects must test their blood sugar twice daily and wear a continuous glucose monitor during the three 72-hour study periods. Subjects will be between 40 and 70 years of age and will be recruited from the surrounding community using flyers and public service announcements. Consent will take place in the Department of Nutrition at Loma Linda University by the study investigators. In total, subject participation will last 5 weeks and all meals will be provided during the 3 study periods.

ELIGIBILITY:
Inclusion Criteria:

* adults between age 40 and 70 years with type 2 diabetes
* duration of type 2 diabetes more than 6 months but less than 10 years
* HbA1c 6.0-8.0%
* BMI 25-40 kg/m2
* diet controlled or stable dose of metformin for at least 3 months
* willing to test blood glucose with personal meter twice a day during study test days

Exclusion Criteria:

* using oral hypoglycemic agents or insulin
* history of ischemic heart disease or congestive heart failure
* history of severe diabetic complication (neuropathy, renal failure, stroke)
* taking medication affecting glucose levels (i.e. corticosteroids)
* active infectious disease
* active malignancy
* pregnant or breast feeding woman
* smoker
* history of daily caffeine or alcohol intake
* known allergy to nuts
* lactose or gluten intolerance

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Within-day glucose variability | 3 days
  The primary objective is to evaluate the effect of two isocaloric walnut-enriched meal plans versus a walnut-free ADA meal plan on within-day glucose variability in adults with diabetes by assessing: a) the overall standard deviation (SD) around the sensor glucose calculated for each day and then averaged over the 3-day study periods; b) the mean amplitude of glycemic excursions (MAGE) over the 3-day study periods.

SECONDARY OUTCOMES:
Glucose variability dose response | 3 days
  A secondary objective will be to test for a dose-response effect, i.e. the more walnuts (full-dose versus half-dose) the lower the glucose variability.
Dose response to between-day glycemic variability | 3 days
  The effect of the three isocaloric ADA meal plans (full-dose, half-dose, walnut free) on the mean of the daily differences(MODD) will be recorded as a measure of between-day glycemic variability
Glucose levels by meal | 3 days
  Glucose levels will be measured before and after breakfast, lunch and dinner for each of the three isocaloric ADA meal plans (full-dose, half-dose, walnut free)
Mean glucose of sensor range | 3 days
  The mean of the glucose for the range captured on each sensor (sensor maximal glucose level minus minimal glucose level will be recorded
Duration of hypoglycemia | 3 days
  The duration of hypoglycemia will be measured as hours per day for each of the three isocaloric ADA meal plans (full-dose, half-dose, walnut free)
Duration of hyperglycemia | 3 days
  The duration of hyperglycemia will be measured as hours per day for each of the three isocaloric ADA meal plans (full-dose, half-dose, walnut free)
Net glycemia at 2 hours | 3 days
  The continuous overall net glycemic action will be measured at 2 hour intervals
Net glycemia at 4 hours | 3 days
  The continuous overall net glycemic action will be measured at 4 hour intervals

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Wien, DrPH, RD, Principal Investigator — Assistant Professor
Locations (1):
- Loma Linda University, Nichol Hall, Loma Linda, California, United States